CLINICAL TRIAL: NCT07195188
Title: The Effect of Game-based Education on Adherence to Treatment and Anxiety Level in Type 2 Diabetics Started on Insulin Therapy
Brief Title: Game-Based Education and Treatment Adherence in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Tinaztepe University (Other)
Collaborators: Usak State Hospital (Other)
Responsible Party: Principal Investigator, gönül düzgün, assistant profesor, Izmir Tinaztepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 352-352-10
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Diabete Mellitus
Keywords: Type 2 Diabetes, Insulin Therapy, Game-Based Education, Treatment Adherence, Anxiety, Randomized Controlled Study, Nursing Education, Patient Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Treatment Adherence and Compliance; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-Based Education (Experimental): Arm Description:
  Participants in this group will receive diabetes education using the "Let's Learn Diabetes" board game. The program consists of four weekly sessions, each lasting two hours, conducted over one month. The sessions aim to improve diabetes knowledge, reduce anxiety, and increase adherence to insulin therapy.
  Interventions: Behavioral: "Let's Learn Diabetes" Game-Based Education
- Traditional Diabetes Education (Active Comparator): Participants in the control group will receive standard diabetes education through traditional lecture-based presentations. The education schedule matches the experimental group with four weekly sessions, each lasting two hours, over one month.
  Interventions: Behavioral: Traditional Diabetes Education

INTERVENTIONS:
Behavioral: "Let's Learn Diabetes" Game-Based Education — Participants in the experimental group will receive diabetes education using the "Let's Learn Diabetes" board game. The program consists of four weekly sessions, each lasting two hours, over one month. The intervention is designed to improve diabetes knowledge, reduce anxiety, and enhance treatment adherence among patients with Type 2 Diabetes Mellitus on insulin therapy.
  Arms: Game-Based Education
Behavioral: Traditional Diabetes Education — Participants in the control group will receive standard diabetes education through traditional lecture-based presentations. The education schedule matches the experimental group with four weekly sessions, each lasting two hours, over one month.
  Arms: Traditional Diabetes Education

SUMMARY:
The goal of this clinical trial is to learn if an education program can help lower anxiety and improve treatment follow-up in adults with type 2 diabetes. The main questions it aims to answer are:

Does attending the education program lower anxiety levels?

Does it help people better follow their diabetes treatment plan?

Researchers will compare two groups:

Education group: Participants who attend the program.

Control group: Participants who do not attend the program.

Participants will:

Be randomly assigned to either the education group or the control group.

Attend four weekly sessions, each lasting two hours, over one month (education group only).

Complete surveys before and after the program, including the Beck Anxiety Scale (to measure anxiety) and the Patient Compliance Scale for Type 2 Diabetes Mellitus Treatment (to measure treatment follow-up).

DETAILED DESCRIPTION:
Study Type: This is a clinical trial that tests a diabetes education program. Number of Participants: A total of 72 people participated in the study

Group Assignment: Participants were randomly assigned to one of two groups:

Game-Based Education Group Traditional Education Group Study Model: Both groups were given diabetes education simultaneously, but through different methods Blinding: This was an open-label study in which both the researchers and the participants were aware of the type of education they received

Main Goal: To test whether a game-based education program can:

Improve how well people follow their diabetes treatment plan Lower anxiety levels in people recently starting insulin therapy Groups and Interventions

1. Game-Based Education Group (Experimental Group) Intervention: "Let's Learn Diabetes" Board Game

   Description:

   Participants received diabetes education through an interactive, game-based program.

   The program consisted of four weekly sessions, each lasting two hours, over the course of one month

   The sessions involved group play to help participants:

   Improve their knowledge about diabetes Reduce anxiety related to diabetes care Follow their treatment plan more closely
2. Traditional Education Group (Control Group) Intervention: Standard Diabetes Education via Lecture

Description:

Participants received standard education using lecture-style presentations. The schedule was the same as the game-based group: four weekly sessions, each two hours long.

Study Outcomes

Researchers measured two main outcomes before the study and one month after the last session:

Treatment Adherence How well participants followed their treatment plan. Measured using the Patient Compliance Scale for Type 2 Diabetes Mellitus Treatment (a survey that asks questions about treatment follow-up).

Anxiety Levels How anxious participants felt about their condition and treatment. Measured using the Beck Anxiety Scale (a survey that measures anxiety).

Who Could Join the Study

Participants were eligible if they:

Had a diagnosis of type 2 diabetes. Started insulin treatment within the past three months. Were 18 years or older. Could read and understand Turkish, since the program was in Turkish. Were willing to sign a consent form and take part in all study activities.

Participants were NOT eligible if they:

Had cognitive problems, severe psychiatric disorders, or dementia that would make participation difficult.

Had severe diabetes-related complications, such as diabetic ketoacidosis or advanced kidney failure.

Had completed a structured diabetes education program in the last six months. Had any other condition that researchers believed would make participation unsafe or inappropriate.

Timeline Study Start Date: April 2024 Final Data Collection Date: October 2024

Program Duration per Participant:

4 weeks total - one two-hour session each week. A follow-up check was done one month after the final session.

Location

The study was carried out at:

Uşak Training and Research Hospital, Diabetes Education Unit and Diabetes School, Uşak, Turkey.

ELIGIBILITY:
nclusion Criteria:

Age at diagnosis of diabetes is at least 1 year.

The maximum duration of insulin treatment initiation is 3 months.

Not having any mental problems.

Between the ages of 40 and 65 years.

Volunteering to participate in the study.

Exclusion Criteria:

Age at diagnosis of diabetes is recent or less than 1 year.

Being on insulin therapy for more than three months.

Mental or psychological comorbidity.

Not within the target age range, under 40 years or over 65 years.

Refusing to participate in the research.

Not attending one or more of the four training sessions during the research process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Treatment Compliance Levels | Pre-intervention and Post-intervention (After 1 Month of Training)
  For Treatment Compliance: The level of compliance among individuals undergoing diabetes-to-diabetes treatment was determined using the Patient Compliance Scale for Type 2 Diabetes Treatment, a 30-item, five-point Likert-type scale. A low total score indicates high patient compliance.
  For Anxiety: "Anxiety levels of individuals with diabetes were determined using the Beck Anxiety Scale (BAS), a 21-item, four-point Likert-type self-report scale. Higher scores indicate more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül düzgün, phd, Study Director — Izmir Tinaztepe University
Locations (1):
- Uşak Eğitim Ve Araştırma Hastanesi, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT07195188/Prot_SAP_000.pdf